CLINICAL TRIAL: NCT04041921
Title: A Multicenter, Prospective, Real World Observational Study for Chronic Total Occlusion
Brief Title: Chronic Total Occlusion Registry
Acronym: IRIS CTO
Status: Terminated | Type: Observational
Why Stopped: The purpose of this study is no longer maintained
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor,University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: CVRF2009-06
Record Dates: First submitted 2019-07-25; First posted 2019-08-01 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Coronary Occlusion; Coronary Artery Stenosis; Coronary Stenosis
Keywords: CTO; PCI; CABG; Medical treatment; Decision CTO
MeSH Terms: conditions — Coronary Occlusion; Coronary Stenosis | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic coronary occlusion patients: ≥3 months chronic total occlusion on coronary angiography
  Interventions: Procedure: Percutaneous coronary intervention; Procedure: Coronary Artery Bypass Grafting; Drug: Medical treatment

INTERVENTIONS:
Procedure: Percutaneous coronary intervention
Procedure: Coronary Artery Bypass Grafting
Drug: Medical treatment

SUMMARY:
This study evaluated the long-term outcome of patients with chronic total occlusion treated with percutaneous coronary intervention, medical treatment or coronary artery bypass grafting.

DETAILED DESCRIPTION:
This study is connected with Decision-CTO trial(NCT01078051). Randomized subjects and registry group subjects from Decision-CTO trial continue 10 years follow-up on this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angina or silent ischemia and documented ischemia
* Patients with De novo chronic coronary occlusion ≥ 3months and reference diameter ≥ 2.5 mm on coronary angiography
* Age > 18 years

Exclusion Criteria:

* Refuse to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with De novo chronic coronary occlusion ≥ 3months and reference diameter ≥ 2.5 mm on coronary angiography
Sampling Method: Probability Sample
Enrollment: 4006 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Composite event of all cause death, myocardial infarction, stroke or all kinds of repeat revascularization | 10 years

SECONDARY OUTCOMES:
Event rate of all cause death | 10 years
Event rate of acute myocardial infarction | 10 years
Event rate of stroke | 10 years
Event rate of repeat revascularization | 10 years
Event rate of rehospitalization due to acute coronary syndrome | 10 years
The rate change of left ventricular ejection fraction | 10 years
Composite event of death, myocardial, stroke or repeat revascularization | 5 years
Composite event of death, myocardial, stroke or repeat revascularization | 10 years
Event rate of Procedural success | 5 days
  Procedural success is defined as < 30% final stenosis and the absence of in-hospital event including death, Q-wave myocardial infarction or urgent repeat revascularization.

CONTACTS AND LOCATIONS:
Locations (19):
- South Korea (19):
  - SAM hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - ChonBuk National University Hospital, Jeonju
  - Dong-A Medical Center, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Bundang CHA Hospital, Seongnam
  - Asan Medical Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided